CLINICAL TRIAL: NCT03002935
Title: A Phase I Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Orally Administered BPM31510 in Healthy Subjects
Brief Title: A Safety Study of Orally Administered BPM31510 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP 0312-02
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BPM31510 Oral Nanosuspension 4% (Experimental): Study subjects will self-administer 80 mL (4 vials of 20 mL) of oral BPM31510 (Ubidecarenone, USP; 40 mg/mL) nano-suspension 3 times daily every 4 to 6 hours for a total daily dose 9600 mg/day of BPM31510 for 14 consecutive days. The last study dose (morning dose only) is administered at the clinic on Day 15.
  Interventions: Drug: BPM31510 Oral Nanosuspension 4%

INTERVENTIONS:
Drug: BPM31510 Oral Nanosuspension 4% — Oral nanosuspension formulation of BPM31510 (ubidecarenone, USP)
  Other Names: Coenzyme Q10, CoQ10, ubidecarenone

SUMMARY:
This is an open-label, Phase I study of the bioavailability and safety of BPM31510 administered orally in healthy subjects dosed 3 times daily for 14 days. The last study dose is administered on Day 15 (one morning dose only). The study will consist of 25 subjects.

DETAILED DESCRIPTION:
Study subjects will be admitted to the clinic on Day -1. All subjects will self-administer the Day 1 doses of study drug under supervision of the clinic staff. Doses of 3200 mg will be administered three times per day before meals.

Dosing will continue for an additional 14 days on an outpatient basis with Day 5 morning dose and the last study dose on Day 15 to be administered at the clinic (one morning dose, is given on Day 15).

On Days 1, 2, 5 and 15, pharmacokinetic (PK) and pharmacodynamics (PD) sampling will be performed 30 minutes prior to the first dose, and 0.5, 1, 2, and 4 hours after the first dose at all visits with an additional PK draw on Day 1 at 0.5, 1, 2, and 4 after the second dose. Urine for PK/PD will be collected pre-dose on Day 1, Day 2, Day 5 and Day 15. At all visits (on Days 1, 2, 5 and at the final dose on Day 15), samples will be collected for chemistry, Complete Blood Count (CBC), International normalized ratio (INR), prothrombin time (PT), partial thromboplastin time (PTT), cholesterol, low density lipoprotein (LDL), and high density lipoprotein (HDL), and vitamin K level. Blood samples for PK/PD will be collected 30 minutes prior to the morning dose on Day 5 and Day 15 and also at 0.5, 1, 2, and 4 hours after dosing. Lab samples (chemistry, etc.), will also be drawn at the time of the first PK/PD draw on Day 5 and Day 15.

A phone interview will be conducted no fewer than 25 days and no more than 35 days after the last dose on Day 15 to collect information on concomitant medications and adverse events Graded using Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age >18 years
* Body mass index (BMI)≥19 and ≤30
* Good health conditions or without significant illness, by judgment of a legally qualified professional, according to the following evaluations: medical history, physical examination, vital signs, electrocardiogram (ECG), and screening or baseline hematology and clinical chemistry measures.
* Subjects of child bearing potential must agree to use one of the accepted methods of contraception (listed below) during the trial (including the screening period prior to receiving trial medication), at least until return of menstruation after stopping the trial medication.

  * condom (male or female) with spermicide
  * diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * hormonal contraception and condom (male or female)
* Female subjects must have a negative pregnancy test result at screening and Day-1
* PT/PTT/INR within normal limits
* Vitamin K levels within normal limits
* Capable of understanding and complying with the protocol and signing informed consent

Exclusion Criteria:

* Pregnant or lactating female subjects
* Known hypersensitivity to the study drug (Coenzyme Q10) or to compounds chemically related
* History or presence of hepatic or gastrointestinal illnesses, or other condition that interferes with the drug's absorption, distribution, excretion or metabolism
* History of hepatic, renal, pulmonary, gastrointestinal, epileptic, hematologic or psychiatric illness
* Hypotension or hypertension of any etiologic that needs pharmacologic treatment
* History of or existing coagulopathy
* History of myocardial infarction, angina, and/or heart insufficiency
* Non-recommended electrocardiographic findings, according to investigator criteria
* Results of the laboratory exams out of normal range unless that they are considered as clinically irrelevant by the investigator
* Subject is a smoker
* Subject ingests more than 5 cups of coffee or tea a day
* History of alcohol or drug abuse
* History of serious adverse reactions or hypersensitivity to any drug
* On-going regular use of oral prescription drugs, with the exception of oral contraceptives
* Hospitalization for any reason within 8 weeks prior to study dosing
* Participation in any experimental study or ingested any experimental drug within 30 days preceding study
* Donation or loss of 450 mL or more of blood within the 3 months prior to Screening/Baseline
* Subject consumed alcohol 48 hours prior to the baseline measurements of the study
* Subject reports history of human immunodeficiency virus
* Currently using coenzyme Q10 over-the-counter products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Days 1, 2, 5, 15; baseline pre-dosing concentrations
  Pharmacokinetic (PK) samples collected to establish oral bioavailability.
Area under the plasma concentration curve (AUC0-4) | Days 1, 2, 5, 15; baseline pre-dosing concentrations
  Pharmacokinetic (PK) samples collected to establish oral bioavailability.

SECONDARY OUTCOMES:
Number of study subjects with adverse events | Baseline to 25-35 days after the end of dosing
  A follow-up phone interview with each study subject will occur 25 to 35 days after the end of dosing to measure the number of adverse events that have occurred.
C-reactive protein measurement | Days 1, 2, 5, 15
Cholesterol measurement | Days 1, 2, 5, 15
Low density lipoprotein (LDL) measurement | Days 1, 2, 5, 15
High density lipoprotein (HDL) measurement | Days 1, 2, 5, 15

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Shenouda, MD, Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs Inc., Eatontown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No